CLINICAL TRIAL: NCT07009067
Title: Safety and Efficacy of Cardiac Rehabilitation With Exercise in Patients With Type-B Aortic Dissection and Intervention: Pilot Study
Brief Title: Safety and Efficacy of Exercise in Type-B Aortic Dissection
Acronym: SECRET-Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Huan Ma, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025-203
Record Dates: First submitted 2025-04-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Type B Aortic Dissection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation Group (Experimental)
  Interventions: Behavioral: Exercise-based Cardiac Rehabilitation
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Exercise-based Cardiac Rehabilitation — Participated will receive 36 individualized Exercise-based Cardiac Rehabilitation after enrollment in our Cardiac Rehabilitation Center.
  Arms: Rehabilitation Group

SUMMARY:
This is a pilot study. The goal of this clinical trial is to evaluate the safety and efficacy of exercise-based cardiac rehabilitation in patients with Type-B Aortic dissection or intramural hematoma or penetrating ulcer and received endovascular repair. The main questions it aims to answer are:

• Is exercise-based cardiac rehabilitation safe among these patients? Participants will be randomly assigned to receive usual care plus exercise-based cardiac rehabilitation (guided exercise for 3 months in rehabilitation center) or usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a previous diagnosis of type B aortic dissection or intramural hematoma or penetrating ulcer, who underwent endovascular aortic repair (EVAR) or EVAR + supra-aortic shunt surgery for more than 1 month, and no related complications (such as endoleak, stent thrombosis, dissection progression, etc.) were found in the postoperative aortic CTA;
* Able to independently carry out basic daily life activities, participants must be able to complete the baseline assessment and start the designated treatment;
* Patients voluntarily participate in this study, sign the written informed consent, and are willing to cooperate with the follow-up;

Exclusion Criteria:

* Acute myocardial infarction occurred 1 month ago;
* Combined with severe aortic stenosis or regurgitation;
* Combined with ascending aortic aneurysm or dissection;
* Acute heart failure occurred 2 weeks ago;
* Combined with severe hypertrophic obstructive cardiomyopathy;
* Chronic renal failure stage 5, which is defined as glomerular filtration rate <15ml/(min·1.73m2) or dialysis;
* During the screening examination, the patient's alanine aminotransferase or aspartate aminotransferase is greater than or equal to 5 times the upper limit of the normal value specified by our center;
* Patients with any medical history that may affect compliance with the program;
* Patients with severe language, mental or physical disabilities who are unable to participate in the program;
* Pregnant or lactating women, or those with fertility who are unwilling/unable to take effective contraceptive measures;
* Patients participating in other interventional clinical trials;
* Patients with long-term high-intensity exercise habits;
* Patients who are judged by the researchers to be unsuitable for participation in this study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events during exercise | 3 months
  Rates of blood pressure increase ≥ 180/100 mmHg, new myocardial ischemia, and new arrhythmia during exercise; rates of dyspnea, palpitations, dizziness/syncope during exercise; and new chest pain/low back pain or worsening chest pain/low back pain
Aortic diameter | 3 months
  The difference of aortic diameter before and after after 3-month intervention in mm.
Progression of dissection | 3 months
  Increase in the number of aorta and its main branches involved in the dissection, the length of a single vessel dissection increases by more than 10 mm, or part of the dissected vessel ruptures
Endoleak | 3 months
  Incidence of new endoleak after 3-month intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No